CLINICAL TRIAL: NCT04419402
Title: ENZA-p: A Randomised Phase II Trial Using PSMA as a Therapeutic Agent and Prognostic Indicator in Men With Metastatic Castration-resistant Prostate Cancer Treated With Enzalutamide (ANZUP 1901)
Brief Title: Enzalutamide With Lu PSMA-617 Versus Enzalutamide Alone in Men With Metastatic Castration-resistant Prostate Cancer
Acronym: ENZA-p
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: National Health and Medical Research Council, Clinical Trials Centre (Unknown); Prostate Cancer Research Alliance (Unknown); Endocyte (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1901
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lu-PSMA + Enzalutamide (Experimental): Lu-PSMA - 7.5 GBq (± 10%): doses 1 and 2 (Days 15 and 57). Doses 3 and 4 (Days 113 and 169) will be given following result of PSMA PET/CT scans at Day 92.
  Enzalumatide - 160 mg (four 40 mg capsules): daily until participant is no longer clinically benefiting, or experiences unacceptable toxicity.
  Interventions: Drug: Lu-PSMA; Drug: Enzalutamide
- Enzalutamide (Active Comparator): Enzalutamide - 160 mg (four 40 mg capsules): daily until participant is no longer clinically benefiting, or experiences unacceptable toxicity.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Lu-PSMA — Patients will be given 7.5 GBq of Lu-PSMA in 4 doses. Dose 1 and 2 on Days 15 and 57. Doses 3 and 4 (Days 113 and 169) will be given following result of 68Ga-PSMA PET/CT at Day 92.
  Treatment administered every 6 weeks, x 4 cycles.
  Other Names: 177Lutetium -PSMA 617 also referred to as 177Lu-PSMA
  Arms: Lu-PSMA + Enzalutamide
Drug: Enzalutamide — 160 mg (four 40 mg capsules) daily.
  Other Names: Xtandi

SUMMARY:
This phase 2 randomised clinical trial will investigate the activity and safety of adding Lu-PSMA to enzalutamide in patients with metastatic castrate resistant prostate cancer (mCRPC) not previously treated with chemotherapy.

DETAILED DESCRIPTION:
This is an open label, randomised, stratified, 2-arm, multicentre phase 2 clinical trial recruiting 160 participants over 12 months and followed until 150 events occurred (approximately another 18 months). Participants will be randomised to enzalutamide or enzalutamide and Lu-PSMA in a 1:1 ratio. A minimisation approach will be used to minimise chance imbalances across the following stratification factors: study site, volume of disease (>20 versus ≤20 sites of disease measured on 68Ga-PSMA PET/CT), prior treatment with early docetaxel for castration- sensitive disease (yes vs no), and prior treatment with early abiraterone for castration-sensitive disease (yes vs no).

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 or older with metastatic adenocarcinoma of the prostate defined by:

   * Documented histopathology of prostate adenocarcinoma (no features of neuroendocrine carcinoma) OR
   * Metastatic disease typical of prostate cancer
2. Castration-resistant prostate cancer (defined as disease progressing despite castration by orchiectomy or ongoing luteinising hormone-releasing hormone agonist or antagonist).
3. Progressive disease with rising PSA defined by PCWG3 criteria (sequence of 2 rising values at a minimum of 1-week intervals) AND PSA ≥ 5 ng/mL.
4. At least 2 of the following risk factors for early treatment failure with enzalutamide:

   * LDH ≥ ULN
   * ALP ≥ ULN
   * Albumin <35 g/L
   * De novo metastatic disease (M1) at initial diagnosis *
   * <3 years since initial diagnosis
   * >5 bone metastases *
   * Visceral metastases *
   * PSA doubling time <84 days
   * Pain requiring opiates for >14 days
   * Prior treatment with abiraterone * Based on conventional imaging (CT and/or bone scan)
5. Target or non-target lesions according to RECIST 1.1
6. Significant PSMA avidity on 68Ga-PSMA PET/CT, defined as SUVmax >15 at a single site (regardless of lesion size) and SUV max >10 at sites of disease ≥10mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact)
7. ECOG performance status 0-2
8. Adequate renal function:

   - Creatinine clearance ≥ 40mL/ min
9. Adequate liver function:

   * Bilirubin < 1.5 x upper limit of normal (ULN) (or if bilirubin is between 1.5 - 2x ULN, must have a normal conjugated bilirubin)
   * AST or ALT ≤ 2.0 x ULN (or ≤ 5.0 x ULN in the presence of liver metastases)
10. Adequate bone marrow function:

    * Platelets ≥ 100 x109/L
    * Haemoglobin ≥ 90g/L (no red blood cell transfusion in last 4 weeks)
    * Neutrophils > 1.5 x109/L
11. Estimated life expectancy > 12 weeks
12. Study treatment both planned and able to start within 21 days of randomisation
13. Willing and able to comply with all study requirements (including both treatments: enzalutamide and Lu-PSMA), and all required study assessments
14. Signed, written, informed consent

Exclusion Criteria:

1. Prostate cancer with known significant sarcomatoid, or spindle cell, or neuroendocrine small cell components, or metastasis of other cancer to the prostate
2. 68Ga-PSMA PET/CT SUVmax < 10 at a site of measurable disease > 10mm
3. Prior treatment with enzalutamide, darolutamide, or apalutamide. Prior treatment with abiraterone is allowed.
4. Prior treatment with any PSMA-targeted radiotherapy
5. Prior chemotherapy for mCRPC. Prior docetaxel in castration-sensitive setting is permitted
6. History of another malignancy within 5 years prior to randomisation except for non-melanomatous carcinoma of the skin; or, adequately treated, non-muscle-invasive urothelial carcinoma of the bladder (i.e. Tis, Ta and low grade T1 tumours)
7. Concurrent illness, including severe infection that may jeopardise the ability of the participant to undergo the procedures outlined in this protocol with reasonable safety
8. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse
9. Men in sexual relationships with women of reproductive potential who are not willing/able to use medically acceptable forms of barrier contraception
10. History of:

    1. seizure or any condition that may predispose to seizure (e.g. prior cortical stroke or significant brain trauma)
    2. loss of consciousness or transient ischemic attack within 12 months of randomization
    3. significant cardiovascular disease within the last 3 months: including myocardial infarction, unstable angina, congestive heart failure (NYHA grade II or greater, see Appendix 4), ongoing arrhythmias of Grade > 2, thromboembolic events (e.g. deep vein thrombosis, pulmonary embolism). Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with mCRPC not previously treated with docetaxel for castration-resistant disease, suitable for treatment with enzalutamide and Lu-PSMA.
Enrollment: 162 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) Progression-Free Survival | Date of randomisation to the date of first evidence of PSA progression - assessed up to study completion, approximately 4 years from recruitment.
  PSA progression is defined as a rise in PSA by more than or equal to 25% AND more than or equal to 2 ng/mL above the nadir (lowest PSA point). This needs to be confirmed by a repeat PSA performed at least 3 weeks later.

SECONDARY OUTCOMES:
Radiographic Progression-Free Survival | Date of randomisation to the date of first evidence of radiographic progression on imaging. Assessed every 12 weeks through study completion, approximately 4 years from start of recruitment.
  Radiographic progression-free survival is defined as the interval from the date of randomisation to the date of first evidence of radiographic progression on imaging, or the date of last known follow-up without progression.
Prostate Specific Antigen (PSA) response rate | Date of randomisation through study completion, approximately 4 years from start of recruitment. Early rises in PSA prior to 12 weeks will be disregarded in determining PSA response
  PSA response rate is defined as the proportion of participants in each group with a PSA reduction of 50% or more from baseline.
Pain response and Progression-Free Survival | Date of randomisation through study completion, approximately 4 years from start of recruitment
  Pain is measured using the McGill-Melzack Present Pain Intensity scale (PPI). Pain Response is defined as a reduction of 2 or more points for participants with a baseline PPI score of 2 or more. Pain progression is defined as and an increase of 1 or more points in the nadir PPI score.
  Pain Response is defined as a reduction of 2 or more points for participants with a baseline PPI score of 2 or more.
  Pain progression is defined as and an increase of 1 or more points in the nadir PPI score.
Clinical Progression-Free Survival | Date of randomisation to the date of first clinical evidence of disease progression or death from any cause. Assessed up to study completion approximately 4 years from recruitment.
  Clinical progression is defined by progression on imaging, development of symptoms attributable to cancer progression, the need for radiotherapy to new metastases or initiation of other anticancer treatment for prostate cancer.
Aspects of Health-related Quality of life (HRQL) | Assessed every 4-6 weeks, through study completion, approximately 4 years from recruitment.
  The European Organisation for Research and Treatment of Cancer (EORTC) core quality of life questionnaire includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), and a global health and quality-of-life scale to assess HRQL in cancer patients. The Patient DATA form is a simple, multi-item quality of life instrument based on 11-point numeric rating scales for a range of relevant symptoms and functions. It combines cancer specific items from the UBQ-C, GLQ-8 and LASA cancer-specific quality of life instruments. The Fear of Cancer Progression form is a short questionnaire assessing possible future concerns related to the participant's illness.
Frequency and Severity of Adverse Events | Through study completion, approximately 4 years from recruitment.
  The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 will be used to classify and grade the intensity of adverse events during study treatment.

OTHER OUTCOMES:
Overall Survival | Through study completion, approximately 4 years from recruitment.
  Overall survival is defined as the interval from date of randomisation to the date of death from any cause, or the date of last known follow-up alive.
Resource Use and Incremental Cost-effectiveness | Through study completion, approximately 4 years from recruitment.
  Information on health-care resource use will be combined with information on overall survival and quality of life to estimate the value associated with the addition of Lu-PSMA to enzalutamide in terms of the cost per Quality adjusted life year (QALY).
Association between Clinical Outcomes and Imaging Analyses at Baseline and During Treatment | Through study completion, approximately 4 years from recruitment.
  A variety of methods to develop, validate and compare predictive and prognostic biomarkers for both enzalutamide treatment and enzalutamide and Lu-PSMA therapy. These include but are not limited to analyses of: 1. associations of screening whole body quantitative parameters on 68Ga-PSMA PET/CT and 18F FDG PET/CT; 2. association between the change on whole body quantitative PET parameters; 3. using the 68Ga-PSMA PET/CT at Day 92, assessment of quantitative whole body PET findings will help determine the proportion of men with persistent PSMA avid disease volume in those undergoing either enzalutamide or enzalutamide and Lu-PSMA treatments; 4. a visual scoring system for both 68Ga-PSMA PET/CT and 18F FDG PET/ CT to evaluate and validate its use in treatment response; 5. QTBI (Quantitative total body imaging) heterogeneity assessment.
Association between Clinical Outcomes and Possible Prognostic/Predictive Biomarkers (tissue and circulating) including CTCs and ctDNA | Through to study completion, approximately 4 years from recruitment.
  Translational research will include identifying tissue and circulating biomarkers that are prognostic and/or predictive of response to treatment, safety and resistance to study treatment (associations of biomarkers with clinical outcomes). These include, but are not limited to analyses of: 1. Liquid biopsies: Liquid biopsies will be collected at molecular imaging time points including at baseline, Day 92 and at first progression; 2. CTC: CTCs may be enumerated and analysed at the above time points for a variety of biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Emmett, MBBS, FRACP, Study Chair — St Vincent's Hospital, Sydney
Locations (15):
- Australia (15):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincents Hospital, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Northern Cancer Institute, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Emmett L, Papa N, Subramaniam S, Crumbaker M, Nguyen A, Joshua AM, Sandhu S, Weickhardt A, Lee ST, Ng S, Francis RJ, Goh JC, Pattison DA, Tan TH, Kirkwood ID, Ayati N, Niu C, Hofman MS, Martin AJ, Thomas H, Davis ID, Stockler MR; ENZA-p Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. Prognostic and predictive value of baseline PSMA-PET total tumour volume and SUVmean in metastatic castration-resistant prostate cancer in ENZA-p (ANZUP1901): a substudy from a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2025 Sep;26(9):1168-1177. doi: 10.1016/S1470-2045(25)00339-0. Epub 2025 Jul 30. PMID 40752515
- [Derived] Emmett L, Subramaniam S, Crumbaker M, Joshua AM, Sandhu S, Nguyen A, Weickhardt A, Lee ST, Ng S, Francis RJ, Goh JC, Pattison DA, Tan TH, Kirkwood ID, Gedye C, Rutherford NK, Kumar ASR, Pook D, Ramdave S, Nadebaum DP, Voskoboynik M, Redfern AD, Macdonald W, Krieger L, Schembri G, Chua W, Lin P, Horvath L, Bastick P, Butler P, Zhang AY, McJannett M, Thomas H, Langford A, Hofman MS, Martin AJ, Davis ID, Stockler MR; ENZA-p Trial Investigators; Australian and New Zealand Urogenital and Prostate Cancer Trials Group. Overall survival and quality of life with [177Lu]Lu-PSMA-617 plus enzalutamide versus enzalutamide alone in metastatic castration-resistant prostate cancer (ENZA-p): secondary outcomes from a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2025 Mar;26(3):291-299. doi: 10.1016/S1470-2045(25)00009-9. Epub 2025 Feb 13. PMID 39956124
- [Derived] Emmett L, Subramaniam S, Crumbaker M, Nguyen A, Joshua AM, Weickhardt A, Lee ST, Ng S, Francis RJ, Goh JC, Pattison DA, Tan TH, Kirkwood ID, Gedye C, Rutherford NK, Sandhu S, Kumar AR, Pook D, Ramdave S, Nadebaum DP, Voskoboynik M, Redfern AD, Macdonald W, Krieger L, Schembri G, Chua W, Lin P, Horvath L, Bastick P, Butler P, Zhang AY, Yip S, Thomas H, Langford A, Hofman MS, McJannett M, Martin AJ, Stockler MR, Davis ID; ENZA-p Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. [177Lu]Lu-PSMA-617 plus enzalutamide in patients with metastatic castration-resistant prostate cancer (ENZA-p): an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2024 May;25(5):563-571. doi: 10.1016/S1470-2045(24)00135-9. Epub 2024 Apr 12. PMID 38621400
- See also: Description: Sponsor's website — http://www.anzup.org.au